CLINICAL TRIAL: NCT01607554
Title: A Pilot, Non-Randomized Phase II Protocol of Irinotecan for Patients With Previously Treated, Advanced, Non-Small Cell Lung Cancer With High ISG 15 Expression
Brief Title: Irinotecan for Previously Treated, Advanced, Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inadequate enrollment (2 subjects in 4 years)
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: University of New Mexico Cancer Center (Other); Lovelace Respiratory Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1201; NCI-2012-01531 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-05-09; First posted 2012-05-30 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung; non small cell; NSCLC; Irinotecan
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan (Experimental): The starting dose of irinotecan for the study is 180 mg/m2, given intravenously every 14 days. Each 14 day period will constitute one cycle of treatment.
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — 180 mg/m2 Irinotecan intravenously over 60 minutes on day 1 of each cycle
  Pre-medication for irinotecan: palonosetron 0.25 mg and dexamethasone 8 - 16 mg, both administered intravenously. Atropine 0.25 - 0.5 mg subcutaneously or IV is at the discretion of the treating physician
  Other Names: Camptosar; Campto

SUMMARY:
Certain genetic factors can affect a patient's potential sensitivity to therapeutic drugs and other agents. There is a factor called ISG15 which might help doctors better identify patients with advanced non-small cell lung cancer (NSCLC) whose tumors may be more sensitive to the drug called Irinotecan. This factor is elevated in roughly 30% of NSCLC cases. Irinotecan is an agent that inhibits the enzyme called topoisomerase I that is involved in cell growth, and it has been FDA approved for 17 years for another type of cancer.

DETAILED DESCRIPTION:
The goal of this trial is to demonstrate the potential clinical benefit of targeted irinotecan chemotherapy in NSCLC patients whose tumors display a specific phenotype that is associated with increased sensitivity to this drug, ISG15H.

ELIGIBILITY:
Inclusion Criteria:

-INCLUSION:

18 years of age or older Have received prior chemotherapy for histologically proven advanced non-small cell lung cancer, up to 3 prior treatments Tumors display high ISG15 (ISG15H) at screening Life expectancy of at least 12 weeks ECOG/Zubrod performance status of 0-2 Provide informed consent permission to participate

Adequate bone marrow function as follows:

1. Absolute neutrophil count of greater than or equal to 1,500 or cells/mm3, and 2) Platelet count greater than or equal to 100,000/mm3 and 3) Absence of a regular red blood cell transfusion requirement

Adequate hepatic function with:

1. Total bilirubin less than or equal to 4.0 mg/dl, and
2. SGOT or SGPT less than or equal to four times ULN

Adequate renal function as defined by:

1) Serum creatinine less than or equal to 1.5 x ULN

Exclusion Criteria:

Symptomatic brain metastases

Pregnant women or nursing mothers

Patients of child bearing potential must use adequate contraception.

May not be receiving other concurrent chemotherapy or radiation therapy

Severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections

Previous hypersensitivity reaction to camptothecins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J Edelman, MD, Principal Investigator — UNM Cancer Center; Mathewos Tessema, PhD, Principal Investigator — Lovelace Respiratory Research Institute
Locations (3):
- United States (3):
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Cancer Center, an NCI Designated Cancer Center — http://cancer.unm.edu/
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan: The starting dose of irinotecan for the study is 180 mg/m2, given intravenously every 14 days. Each 14 day period will constitute one cycle of treatment.
  Irinotecan: 180 mg/m2 Irinotecan intravenously over 60 minutes on day 1 of each cycle
  Pre-medication for irinotecan: palonosetron 0.25 mg and dexamethasone 8 - 16 mg, both administered intravenously. Atropine 0.25 - 0.5 mg subcutaneously or IV is at the discretion of the treating physician
Period: Overall Study
Arm/Group | Irinotecan
Started | 2
Completed | 0
Not Completed | 2
Not completed — Disease progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Change in tumor size will be measured by CT scan using RECIST criteria.
Time Frame: 8 weeks
Population: Both participants experienced an increase in tumor size between the time of the baseline CT scan and the first study CT scan. There will be no publication or further data analysis, as the study was terminated early due to low enrollment (2) and the original PI has left employment with the institution.
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression will be measured from the time of first treatment until there is evidence of progressive disease or death, from the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 100 months. Death will be treated as a progression event.
Time Frame: Up to 100 months
Population: No data were collected on this outcome measure. There will be no publication or data analysis, as the study was terminated early due to low enrollment (2) and the original PI has left employment with the institution.
Arm/Group | Irinotecan
Number analyzed (Participants) | 0

3. Secondary Outcome: Retrospectively Evaluate the Role of Tumor SULF2 Gene Methylation Status in Treatment Efficacy
Description: Patients who have a loss of SULF2 gene expression have a better outcome than those whose tumors express SULF2. High level of ISG15 expression in NSCLC may indicate a subgroup of tumors that may be more sensitive to the cytotoxic effects of irinotecan. In patients who consent to screening, 10 unstained slides of archived diagnostic tissue will be obtained from formalin-fixed, paraffin-embedded specimens and analyzed in the laboratories of our Lovelace Respiratory Research Institute co-investigators.
Time Frame: 1 year
Population: No data was collected for this outcome measure. There will be no publication or data analysis, as the study was terminated early due to low enrollment (2) and the original PI has left employment with the institution.
Arm/Group | Irinotecan
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity of Irinotecan Salvage Chemotherapy
Description: Use blood samples to measure possible 1) Neutropenia, 2) Thrombocytopenia, 3)Diarrhea; 4) Other measures of toxicity other than alopecia, anorexia, and asthenia as listed in the National Cancer Institute Common Toxicity Criteria v. 4.03
Time Frame: 2 days preceding each cycle of therapy
Population: There will be no publication or data analysis, as the study was terminated early due to low enrollment (2) and the original PI has left employment with the institution.
Arm/Group | Irinotecan
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: Up to 100 months
Population: No data were collected for this outcome measure. There will be no publication or data analysis, as the study was terminated early due to low enrollment (2) and the original PI has left employment with the institution.
Arm/Group | Irinotecan
Number analyzed (Participants) | 0

6. Secondary Outcome: Median Duration of Response
Time Frame: Up to 100 months
Population: as for outcome 5
Arm/Group | Irinotecan
Number analyzed (Participants) | 0

7. Secondary Outcome: Median Overall Survival (OS)
Time Frame: 100 months
Population: as for outcome 5
Arm/Group | Irinotecan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Irinotecan
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan (N=2)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan (N=2)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Alopecia (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (3)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Alkaline phosphatase increased (Hepatobiliary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (3)
Anorexia (General disorders) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Renal and urinary disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (4)
Hypoalbuminemia (General disorders) | 2 (4)
Hypokalemia (General disorders) | 1 (1)
Hyponatremia (General disorders) | 1 (1)
Hypophosphatemia (General disorders) | 1 (2)
INR increased (Blood and lymphatic system disorders) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to no subjects analyzed. There will be no publication, as the original PI has left employment with the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No